CLINICAL TRIAL: NCT03035760
Title: A Phase 1 Open Label, Multiple Ascending Dose Study of Oxfendazole in Healthy Adult Volunteers
Brief Title: Multiple Ascending Dose Study of Oxfendazole in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0005; HHSN272201300020I
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2017-07-19

CONDITIONS: Helminthic Infection
Keywords: Helminths; Oxfendazole; Pharmacokinetics; Safety
MeSH Terms: conditions — Trematode Infections | interventions — oxfendazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 (Experimental): 3 mg/kg orally once daily for 5 days (n = 8)
  Interventions: Drug: Oxfendazole
- 2 (Experimental): 7.5 mg/kg orally once daily for 5 days (n = 8)
  Interventions: Drug: Oxfendazole
- 3 (Experimental): 15 mg/kg orally once daily for 5 days (n = 8)
  Interventions: Drug: Oxfendazole
- 4 (Experimental): 3 mg/kg orally, one dose received following a fast (n=6) or high fat meal (n=6) on Day 1 and crossed over to opposite arm to receive drug following high fat meal or fast on Day 8
  Interventions: Drug: Oxfendazole

INTERVENTIONS:
Drug: Oxfendazole — methyl-5 (6)-phenylsulfiyl-2-benzimidazole carbamate, is a broad spectrum benzimidazole antihelminthic. It is the sulphoxide metabolite of fenbendazole.

SUMMARY:
This Phase I study is an open label multiple ascending dose evaluation of the safety and PK of oxfendazole (3, 7.5, or 15 mg/kg) given orally daily to healthy adult men and nonpregnant women aged 18-45 followed by a single dose cross over trial evaluating the safety and pharmacokinetics of a single dose of oxfendazole (3 mg/kg) given following an 8 hour fast or following a high fat meal. The study duration will be approximately 12 months with each subject participation lasting approximately 6 weeks. In the multiple ascending dose evaluation, between 8 and 24 subjects will be enrolled; each dose group will be comprised of eight volunteers. To enhance safety, one sentinel subject will be dosed for five days and monitored for 7 days from the time of the first dose for predefined adverse events. If there are no predefined safety events, a second sentinel subject will be enrolled and followed for a total of 7 days. If there are no predefined safety signals identified for either of these two sentinel subjects, the remaining subjects in the group will be enrolled. After all eight subjects have completed the 10 day follow up period, an electronic safety review of the electronic data will be performed. If none of the predefined safety events have occurred DMID will approve enrollment into the second dose group (7.5 mg/kg oxfendazole daily x 5 days) and will be monitored for a total of 7 days each for predefined adverse events prior to enrolling the remaining subjects in the group. After the 10 day follow up period has been completed for group 2, an electronic safety review will be completed and if no predefined events have occurred two sequential subjects (one at a time with 7 days between each subject) will be enrolled into the third dose group (15 mg/kg oxfendazole daily x 5 days) and will be monitored for a total of 7 days each for predefined safety events prior to enrolling the remaining subjects in the group. In the food effects evaluation, 12 subjects will be enrolled into the single dose cross over group where half of the subjects will initially receive a single dose of 3 mg/kg of oxfendazole following an 8 hour fast and the other half will receive a single dose of 3 mg/kg of oxfendazole following a high fat meal. Subjects will then cross over to receive a single dose following a high fat breakfast or fasting period (water is permitted). All subjects will have received a dose of oxfendazole following both a fasting period and a meal. The primary objectives are: 1) To assess the safety of oxfendazole administered daily for five days; and 2) To assess the safety of oxfendazole administered as a single dose with or without food.

DETAILED DESCRIPTION:
This Phase I study is an open label multiple ascending dose evaluation of the safety and PK of oxfendazole (3, 7.5, or 15 mg/kg) given orally daily to healthy adult men and nonpregnant women aged 18-45 followed by a single dose cross over trial evaluating the safety and pharmacokinetics of a single dose of oxfendazole (3 mg/kg) given following an 8 hour fast or following a high fat meal. The study duration will be approximately 12 months with each subject participation lasting approximately 6 weeks. In the multiple ascending dose evaluation, between 8 and 24 subjects will be enrolled; each dose group will be comprised of eight volunteers. To enhance safety, one sentinel subject will be dosed for five days and monitored for 7 days from the time of the first dose for predefined adverse events. If there are no predefined safety events, a second sentinel subject will be enrolled and followed for a total of 7 days. If there are no predefined safety signals identified for either of these two sentinel subjects, the remaining subjects in the group will be enrolled. After all eight subjects have completed the 10 day follow up period, an electronic safety review of the electronic data will be performed. If none of the predefined safety events have occurred DMID will approve enrollment into the second dose group (7.5 mg/kg oxfendazole daily x 5 days) and will be monitored for a total of 7 days each for predefined adverse events prior to enrolling the remaining subjects in the group. After the 10 day follow up period has been completed for group 2, an electronic safety review will be completed and if no predefined events have occurred two sequential subjects (one at a time with 7 days between each subject) will be enrolled into the third dose group (15 mg/kg oxfendazole daily x 5 days) and will be monitored for a total of 7 days each for predefined safety events prior to enrolling the remaining subjects in the group. In the food effects evaluation, 12 subjects will be enrolled into the single dose cross over group where half of the subjects will initially receive a single dose of 3 mg/kg of oxfendazole following an 8 hour fast and the other half will receive a single dose of 3 mg/kg of oxfendazole following a high fat meal. Subjects will then cross over to receive a single dose following a high fat breakfast or fasting period (water is permitted). All subjects will have received a dose of oxfendazole following both a fasting period and a meal. The primary objectives are: 1) To assess the safety of oxfendazole administered daily for five days; and 2) To assess the safety of oxfendazole administered as a single dose with or without food. The secondary objectives are: 1) To define the multi-dose kinetics of oxfendazole; and 2) To determine the effect of food on the kinetics of oxfendazole.

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females between the ages of 18 and 45 years, inclusive.
2. Women of childbearing potential* must agree to practice adequate contraception** for the 28-day period before Day 0 through 4 months after the last dose of study medication.

   * A woman is considered of childbearing potential unless surgically sterile (tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal (=1 year).

   **Acceptable birth control methods include but are not limited to: abstinence from sexual intercourse with men; monogamous relationship with a vasectomized partner; double-barrier methods (condoms, diaphragms, spermicides); intrauterine devices; and licensed hormonal methods.
3. In good health, as judged by the investigator and determined by vital signs*

   *Temperature < 38°C, heart rate <= 100 bpm and > 50 bpm, systolic blood pressure <= 140 mmHg and > 89 mmHg, diastolic blood pressure <= 90 mmHg and = 60 mm Hg, medical history and a targeted physical examination. BMI >= 18 and <= 35. Athletically trained subjects with a pulse >= 45 may be enrolled at the discretion of the principal investigator or designated licensed clinical investigator. Acceptable screening laboratories: Hemoglobin, white blood cell (WBC) count, neutrophil, and platelet counts, INR and PTT within normal ranges. AST < 44 and ALT < 44 and total bilirubin, creatinine must be equal to or below the upper limit of normal (creatinine values below the normal range are acceptable). Random blood glucose must be <140. Urine dipstick testing must be negative for glucose and negative or trace for protein. The following serology tests must be negative: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody. HIV and hepatitis C viral load PCR testing may be performed for individuals suspected of having indeterminate antibody testing.
4. Male participants must be willing to ensure use of condoms and spermicides for 4 months after the last dose study medication.
5. Provide written informed consent before initiation of any study procedures.
6. Willing to be available for all study-required procedures, and visits for the duration of the study.
7. Individuals must agree to abstain from drug or alcohol use for 48 hours prior to enrollment through day 10 or 14.
8. Able to provide a home phone number, and the name, address, and/or email of a person willing to assist with making contact during the follow-up phase of the study.

Exclusion Criteria:

1. Pregnant women, women who are planning to become pregnant in the next 4 months, or women who are breastfeeding.
2. Body temperature >=100.4°F (>=38.0°C) or acute illness within 3 days before administration of study drug (subject may be rescheduled).
3. Chronic or acute medical disorder*

   * Disorders of the cardiac, pulmonary, liver, kidney, neurologic, gastrointestinal or other system, such that in the opinion of the investigator participation in the study creates additional risk to the subject, or to the validity of the study.
4. Use of chronic systemic medications* *Intermittent use of over the counter medications such as acetaminophen, ibuprofen, cold and sinus medications are permitted for enrollment Topical medications, nasal steroids are permitted throughout the study. Use of prescription medications used less than once per week on average are permitted for enrollment. If the subject has taken a short term prescription medication within the past 30 days (e.g. an antibiotic), they should be postponed from enrollment until 30 days have elapsed since the last dose.
5. Has history of sensitivity to related benzimidazole compounds (e.g., albendazole, mebendazole).
6. A diagnosis of schizophrenia, bipolar disease, or history of hospitalization for a psychiatric condition or previous suicide attempt.
7. A history of treatment for any other psychiatric disorder in the past 3 years.*

   *Past treatment for ADHD does not exclude participants from enrollment as long as the medications have been discontinued for a minimum of 3 months and symptoms are well controlled.
8. Received an experimental agent* within 1 month before administration of study drug or expect to receive an experimental agent during the 10 or 14-day study period.

   *Vaccine, drug, biologic, device, blood product, or medication.
9. Any condition that would, in the opinion of the investigator, interfere with the study.*

   *This includes any condition that would place them at an unacceptable risk of injury, render them unable to meet the requirements of the protocol, or that may interfere with successful completion of the study.
10. A history of heavy alcohol* or illicit drug use**, or history of substance abuse#.

    *On average, greater than 7 alcoholic drinks per week. .

    **Other than occasional marijuana use (less than once per week for the past 60 days is acceptable).

    #Alcohol or illicit drugs within the past 3 years.
11. History of chronic tobacco use in the past 60 days.* *A history of occasional tobacco use (less than 1 pack per week on average) is acceptable. Individuals will be counseled to abstain from use of tobacco and marijuana from screening through day 10 or 14.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Bach T, Galbiati S, Kennedy JK, Deye G, Nomicos EYH, Codd EE, Garcia HH, Horton J, Gilman RH, Gonzalez AE, Winokur P, An G. Pharmacokinetics, Safety, and Tolerability of Oxfendazole in Healthy Adults in an Open-Label Phase 1 Multiple Ascending Dose and Food Effect Study. Antimicrob Agents Chemother. 2020 Oct 20;64(11):e01018-20. doi: 10.1128/AAC.01018-20. Print 2020 Oct 20. PMID 32816721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and non-pregnant females recruited from existing volunteer populations and from the communities at large around the clinical site. Participants were enrolled between 05JUN2017 and 10APR2018.
Groups:
- Arm 1: 3 mg/kg Oxfendazole for 5 Days: Participants received 3 mg/kg oxfendazole orally once daily for 5 days
- Arm 2: 7.5 mg/kg Oxfendazole for 5 Days: Participants received 7.5 mg/kg oxfendazole orally once daily for 5 days
- Arm 3: 15 mg/kg Oxfendazole for 5 Days: Participants received 15 mg/kg oxfendazole orally once daily for 5 days
- Arm 4A: 3 mg/kg Oxfendazole Fasted First, Then High Fat Meal: 3 mg/kg oxfendazole orally, one dose received following a fast on Day 1 and 3 mg/kg oxfendazole following a high fat meal on Day 8
- Arm 4B: 3 mg/kg Oxfendazole High Fat Meal First, Then Fasted: 3 mg/kg oxfendazole orally, one dose received following a high fat meal on Day 1 and 3 mg/kg oxfendazole following a fast on Day 8
Period: First Intervention - 10/7 Days Follow-up
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days | Arm 4A: 3 mg/kg Oxfendazole Fasted First, Then High Fat Meal | Arm 4B: 3 mg/kg Oxfendazole High Fat Meal First, Then Fasted
Started | 8 | 8 | 8 | 6 | 6
Completed | 8 | 8 | 8 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Intervention - 7 Days Follow-up
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days | Arm 4A: 3 mg/kg Oxfendazole Fasted First, Then High Fat Meal | Arm 4B: 3 mg/kg Oxfendazole High Fat Meal First, Then Fasted
Started | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects are included in the analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days | Arm 4A: 3 mg/kg Oxfendazole Fasted First, Then High Fat Meal | Arm 4B: 3 mg/kg Oxfendazole High Fat Meal First, Then Fasted | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 6 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 6 | 6 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (9.1) | 27.1 (6.1) | 30.1 (4.4) | 27.7 (5.6) | 32.2 (9.4) | 29.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 1 | 2 | 11
  Male | 7 | 5 | 4 | 5 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 7 | 8 | 7 | 4 | 6 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 7 | 6 | 6 | 4 | 6 | 29
  More than one race | 0 | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 6 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events (AEs) Related to Oxfendazole for Arms 1, 2, and 3
Description: All adverse events, defined as any untoward medical occurrence regardless of its causal relationship to the study treatment, were collected for 14 days after dosing. The PI then determined relatedness to the study drug. Related was defined as "there is a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event."
Time Frame: Day 1 through Day 10
Population: All participants are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days
Number analyzed (Participants) | 8 | 8 | 8
Participants | 3 | 3 | 1

2. Primary Outcome: Number of Subjects Reporting Adverse Events (AEs) Related to Oxfendazole for Arm 4
Description: as for outcome 1
Time Frame: Day 1 through Day 14
Population: All participants are included in the analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 4: 3 mg/kg Oxfendazole, Post Fast: 3 mg/kg oxfendazole orally, one dose received following a fast on Day 1 or on Day 8
- Arm 4: 3 mg/kg Oxfendazole, Post Fed: 3 mg/kg oxfendazole orally, one dose received following a high fat meal on Day 1 or on Day 8
Arm/Group | Arm 4: 3 mg/kg Oxfendazole, Post Fast | Arm 4: 3 mg/kg Oxfendazole, Post Fed
Number analyzed (Participants) | 12 | 12
Participants | 1 | 2

3. Secondary Outcome: Area Under the Concentration Time-curve for a Single Dosing Interval (AUCtau) of Oxfendazole for Arm 1, 2 and 3
Description: AUCtau was defined as the total area under the concentration-time curve from dosing to the end of the 24-hour dosing interval for Dose 1 and Dose 5. AUCtau was calculated using the Linear Up Log Down calculation method.
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose on day 1 and 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 72, 120 hours post-dose on day 5
Population: All participants are included in the analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days
Number analyzed (Participants) | 8 | 8 | 8
ng•hr/mL
  Dose 1 | 30200 (66.7) | 52500 (73.9) | 71800 (50.7)
  Dose 5 | 38200 (33.1) | 65700 (34.5) | 69600 (28.7)

4. Secondary Outcome: Area Under the Concentration Time-curve to the Time of Last Measured Concentration (AUClast) of Oxfendazole for Arm 4
Description: AUClast was defined as the area under the concentration-time curve from dosing to the time of the last measured concentration of that dosing period greater than the lower limit of quantification of the bioanalytical assay. AUClast was calculated using the Linear Up Log Down calculation method.
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose
Population: All participants are included in the analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Groups:
- Arm 4: 3 mg/kg Oxfendazole, Fed/Fasted: 3 mg/kg oxfendazole orally, one dose received following a fast (n=6) or high fat meal (n=6) on Day 1 and crossed over to opposite arm to receive drug following high fat meal or fast on Day 8
Arm/Group | Arm 4: 3 mg/kg Oxfendazole, Fed/Fasted
Number analyzed (Participants) | 12
ng•hr/mL
  Fed | 58900 (25.5)
  Fasted | 31600 (38.0)

5. Secondary Outcome: Maximum Observed Concentration (Cmax) of Oxfendazole in Plasma for Arms 1, 2, and 3
Description: Cmax is defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: as for outcome 3
Population: All participants are included in the analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days
Number analyzed (Participants) | 8 | 8 | 8
ng/mL
  Dose 1 | 2960 (42.7) | 4160 (59.6) | 5990 (53.1)
  Dose 5 | 3500 (16.3) | 5980 (17.8) | 6000 (28.4)

6. Secondary Outcome: Maximum Observed Concentration (Cmax) of Oxfendazole in Plasma for Arm 4
Description: as for outcome 5
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose
Population: All participants are included in the analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 4: 3 mg/kg Oxfendazole, Fed/Fasted
Number analyzed (Participants) | 12
ng/mL
  Fed | 4500 (19.5)
  Fasted | 3010 (40.9)

7. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Oxfendazole for Arms 1, 2, and 3
Description: The apparent terminal elimination half-life (t1/2) was defined as the time required for the drug concentration to decrease by a factor of one-half in the terminal phase computed from concentrations that were measured using a validated HPLCMS/MS method.
Time Frame: as for outcome 3
Population: All participants are included in the analysis population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days
Number analyzed (Participants) | 8 | 8 | 8
hours
  Dose 1 | 7.98 (1.47) | 8.54 (3.62) | 8.35 (0.48)
  Dose 5 | 9.47 (2.34) | 11.00 (3.39) | 12.00 (2.65)

8. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Oxfendazole for Arm 4
Description: as for outcome 7
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose
Population: All participants are included in the analysis population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 4: 3 mg/kg Oxfendazole, Fed/Fasted
Number analyzed (Participants) | 12
hours
  Fed | 8.05 (0.776)
  Fasted | 7.65 (1.26)

9. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Oxfendazole for Arms 1, 2, and 3
Description: Tmax was defined as the time at which the maximum concentration (Cmax) occurs in plasma computed from concentrations that were measured using a validated HPLCMS/MS method.
Time Frame: as for outcome 3
Population: All participants are included in the analysis population.
Measure: Median (Full Range); unit: hours
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days
Number analyzed (Participants) | 8 | 8 | 8
hours
  Dose 1 | 1.96 [1.83 to 8.55] | 2.02 [0.983 to 8.55] | 2.56 [0.983 to 8.92]
  Dose 5 | 1.92 [1.02 to 3.00] | 2.02 [1.78 to 3.08] | 2.49 [0.917 to 3.02]

10. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Oxfendazole for Arm 4
Description: as for outcome 9
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose
Population: All participants are included in the analysis population.
Measure: Median (Full Range); unit: hours
Arm/Group | Arm 4: 3 mg/kg Oxfendazole, Fed/Fasted
Number analyzed (Participants) | 12
hours
  Fed | 8.9 [3.9 to 11.5]
  Fasted | 1.99 [1 to 2.98]

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of receipt of study drug on Day 1 through the final study visit (approximately 10 or 14 days after receipt of study product).
Arm/Group | Arm 1: 3 mg/kg Oxfendazole for 5 Days | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days | Arm 3: 15 mg/kg Oxfendazole for 5 Days | Arm 4: 3 mg/kg Oxfendazole, Post Fast | Arm 4: 3 mg/kg Oxfendazole, Post Fed
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/8 | 3/8 | 2/8 | 1/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 3 mg/kg Oxfendazole for 5 Days (N=8) | Arm 2: 7.5 mg/kg Oxfendazole for 5 Days (N=8) | Arm 3: 15 mg/kg Oxfendazole for 5 Days (N=8) | Arm 4: 3 mg/kg Oxfendazole, Post Fast (N=12) | Arm 4: 3 mg/kg Oxfendazole, Post Fed (N=12)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vessel Puncture Site Haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngial Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03035760/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT03035760/SAP_001.pdf